CLINICAL TRIAL: NCT03669393
Title: A Phase 2, Open-label, Multi-centre Study to Assess the Efficacy and Safety of Intravitreal THR-317 for the Treatment of Macular Telangiectasia Type 1 (MacTel 1)
Brief Title: A Study to Evaluate THR-317 Treatment for Macular Telangiectasia Type 1 (MacTel 1)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ThromboGenics (Industry)
Responsible Party: Sponsor
Organization: Oxurion (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: THR-317-003; 2017-004010-26 (EudraCT Number)
Record Dates: First submitted 2018-09-10; First posted 2018-09-13 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Retinal Telangiectasis; Idiopathic Juxtafoveal Retinal Telangiectasia
MeSH Terms: conditions — Retinal Telangiectasis; Idiopathic Juxtafoveal Retinal Telangiectasia | interventions — TB-403

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- THR-317 (Experimental)
  Interventions: Drug: THR-317 8mg

INTERVENTIONS:
Drug: THR-317 8mg — 3 intravitreal injections of THR-317 8mg, approximately 1 month apart

SUMMARY:
This study is conducted to evaluate the safety of THR-317 when administered intravitreally and to assess the compound's efficacy in reducing central subfield thickness (CST) and improving best-corrected visual acuity (BCVA) in subjects with macular telangiectasia Type 1 (MacTel 1).

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years or older
* Macular oedema caused by MacTel 1, with CST >300µm on SD-OCT
* Written informed consent obtained from the subject prior to screening procedures

Exclusion Criteria:

* Type 1 or type 2 Diabetes Mellitus
* Concurrent disease in the study eye that could require medical or surgical intervention during the study period for up to 30 days after the last study treatment, or could confound interpretation of the results
* Previous confounding treatments / procedures, or their planned / expected use during the study period for up to 30 days after the last administration of study treatment
* Any active ocular / intraocular infection or inflammation in either eye
* Pregnant or lactating female, or female of child-bearing potential not utilising an adequate form of contraception, or male of reproductive potential not utilising contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2019-11-22 (Actual)

PRIMARY OUTCOMES:
Change from baseline in central subfield thickness (CST), based on spectral domain optical coherence tomography (SD-OCT) | At Day 84 (Month 3)

SECONDARY OUTCOMES:
Change from baseline in CST, based on SD-OCT, by study visit | From baseline to Day 140
Change from baseline in area of cystoid spaces, based on SD-OCT, by study visit | From baseline to Day 140
Change from baseline in best-corrected visual acuity (BCVA), by study visit | From Day 0 to Day 140
Incidence of systemic and ocular adverse events including serious adverse events | From Day 0 to Day 140

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Department, Study Director — Oxurion NV.
Locations (3):
- France (2):
  - Hôpital Lariboisière, Paris
  - Hôpital Cochin, Paris
- Hôpital Ophtalmique Jules-Gonin, Lausanne, Switzerland